CLINICAL TRIAL: NCT02179502
Title: Randomized, Double-blind, Placebo-controlled, Dose-escalation Study for the Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of GLPG1690 in Healthy Male Subjects
Brief Title: First-in-Human Single and Multiple Dose of GLPG1690
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1690-CL-101; 2014-000981-23 (EudraCT Number)
Record Dates: First submitted 2014-06-28; First posted 2014-07-01 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1690; Suspensions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLPG1690 single dose (Experimental): Single oral dose of GLPG1690 suspension or solid formulation - ascending doses
  Interventions: Drug: GLPG1690 single ascending doses
- Placebo single dose (Placebo Comparator): Single oral dose of placebo suspension or solid formulation
  Interventions: Drug: Placebo single ascending doses
- GLPG1690 multiple doses (Experimental): Multiple oral doses of GLPG1690 suspension - ascending doses
  Interventions: Drug: GLPG1690, multiple ascending doses, oral suspension
- Placebo multiple doses (Placebo Comparator): Multiple oral doses of placebo suspension
  Interventions: Drug: Placebo, multiple ascending doses, oral suspension

INTERVENTIONS:
Drug: GLPG1690 single ascending doses — Single dose, oral suspension or solid formulation, starting dose of 20mg escalating up to 1500mg
  Arms: GLPG1690 single dose
Drug: Placebo single ascending doses — Single dose, oral suspension or solid formulation matching placebo
  Arms: Placebo single dose
Drug: GLPG1690, multiple ascending doses, oral suspension — Multiple doses, daily for 14 days, oral suspension, anticipated doses: 300mg to 1000mg
  Arms: GLPG1690 multiple doses
Drug: Placebo, multiple ascending doses, oral suspension — Multiple doses, daily for 14 days, oral suspension matching placebo
  Arms: Placebo multiple doses

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety and tolerability after single ascending oral doses of GLPG1690 given to healthy male subjects, compared to placebo. Also, the safety and tolerability of multiple ascending oral doses of GLPG1690 given to healthy male subjects daily for 14 days compared to placebo, will be evaluated.

Furthermore, during the course of the study after single and multiple oral dose administrations, the amount of GLPG1690 present in the blood and urine (pharmacokinetics) as well as the reduction of biomarker levels by GLPG1690 in plasma samples (pharmacodynamics) will be characterized compared to placebo.

The pharmacokinetics of a solid dosage formulation of GLPG1690 will be compared with those of a liquid dosage formulation of GLPG1690.

Also, the potential of cytochrome P450 (CYP)3A4 induction after repeated dosing with GLPG1690 will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1690 in comparison with placebo after a single and multiple oral dose in healthy subjects in terms of adverse events
Number of subjects with abnormal laboratory parameters | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1690 in comparison with placebo after single and multiple oral dose in healthy subjects in terms of abnormal laboratory parameters
Number of subjects with abnormal vital signs | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1690 in comparison with placebo after a single and multiple oral dose in healthy subjects in terms of abnormal vital signs
Number of subjects with abnormal electrocardiogram | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1690 in comparison with placebo after a single and multiple oral dose in healthy subjects in terms of abnormal electrocardiogram
Number of subjects with abnormal physical examination | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1690 in comparison with placebo after a single and multiple oral dose in healthy subjects in terms of abnormal physical examination

SECONDARY OUTCOMES:
The amount of GLPG1690 in plasma | Between Day 1 predose and 48 hours after the (last) dose
  To characterize the amount of GLPG1690 in plasma over time - pharmacokinetics (PK) - after a single and multiple oral dose in healthy subjects, either as liquid or solid formulation
The amount of GLPG1690 in urine | Between Day 1 predose and 24 hours after the (last) dose
  To characterize the amount of GLPG1690 in urine over time - pharmacokinetics (PK) - after a single and multiple oral dose in healthy subjects, either as liquid or solid formulation
Ratio of 6-b-hydroxycortisol/cortisol in urine | Twelve hours before dosing on Day 1 and Day 14
  To assess the potential of CYP3A4 induction after repeated dosing with GLPG1690 by means of the ratio of 6-b-hydroxycortisol/cortisol in urine
Levels of biomarker in plasma | Day 1 predose up to 48 hours post (last) dose
  To characterize the pharmacodynamics (PD) of GLPG1690 by means of reduction of levels of biomarker by GLPG1690 compared to placebo in plasma after single and multiple oral dose in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] van der Aar E, Desrivot J, Dupont S, Heckmann B, Fieuw A, Stutvoet S, Fagard L, Van de Wal K, Helmer E. Safety, Pharmacokinetics, and Pharmacodynamics of the Autotaxin Inhibitor GLPG1690 in Healthy Subjects: Phase 1 Randomized Trials. J Clin Pharmacol. 2019 Oct;59(10):1366-1378. doi: 10.1002/jcph.1424. Epub 2019 Apr 23. PMID 31012984